CLINICAL TRIAL: NCT04408898
Title: A Phase 2 Pilot Study of ADP-A2M4 in Combination With Pembrolizumab in Subjects With Recurrent or Metastatic Head and Neck Cancer
Brief Title: SPEARHEAD 2 Study in Subjects With Recurrent or Metastatic Head and Neck Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Challenges with recruitment
Sponsor: Adaptimmune (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADP 0044-003
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Head and Neck Cancer
Keywords: Cell Therapy; T-cell Therapy; SPEAR T-Cell; Head and Neck Cancer; MAGE-A4; ADP-A2M4; Immuno-oncology
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADP-A2M4 T cells in combination with pembrolizumab (Experimental)
  Interventions: Genetic: ADP-A2M4 in combination with pembrolizumab.

INTERVENTIONS:
Genetic: ADP-A2M4 in combination with pembrolizumab. — Single infusion of autologous genetically modified ADP-A2M4 Dose: 1.0 x109 to 10x109 transduced cells by a single intravenous infusion Repeat doses of pembrolizumab every 3 weeks. Dose: 200mg

SUMMARY:
This is a study to investigate the efficacy and safety of ADP-A2M4 in combination with pembrolizumab in HLA-A*02 eligible and MAGE-A4 positive subjects with recurrent or metastatic Head and Neck cancer.

ELIGIBILITY:
Key Inclusion Criteria

* Age ≥18 and <75 years
* Diagnosis of head and neck squamous cell carcinoma with metastatic or unresectable, recurrent disease. confirmed by histology cytology.
* Checkpoint inhibitor naïve and indicated for pembrolizumab or currently receiving pembrolizumab (monotherapy). May have received prior platinum containing chemotherapy regimen or checkpoint inhibitor therapy.
* Subjects that have already received pembrolizumab (alone or in combination) and are progressing or have completed immune checkpoint inhibitor therapy for recurrent/metastatic disease, may still be enrolled and will skip Part A of the study.

These subjects will enroll into Part B when manufactured T cells are available.

* Measurable disease according to RECIST v1.1.
* HLA-A*02 positive by central laboratory.
* Tumor shows MAGE-A4 expression confirmed by central laboratory.
* ECOG Performance Status of 0 or 1.
* Left ventricular ejection fraction (LVEF) ≥50%.

Note: other protocol defined Inclusion criteria may apply

Key Exclusion Criteria:

* Positive for any HLA-A*02 allele other than: one of the inclusion alleles, HLA- A*02:07P or HLA-A*02 null alleles
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to fludarabine, cyclophosphamide or other agents used in the study or history of severe hypersensitivity to another monoclonal antibody.
* History of autoimmune or immune mediated disease
* Leptomeningeal disease, carcinomatous meningitis or CNS metastases.
* Other prior malignancy that is not considered by the Investigator to be in complete remission
* Clinically significant cardiovascular disease
* Uncontrolled intercurrent illness
* Active infection with human immunodeficiency virus, hepatitis B virus, hepatitis C virus, or human T cell leukemia virus
* Pregnant or breastfeeding

Note: other protocol defined Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Overall Response Rate (ORR) | 2.5 years
  ORR is defined as the proportion of complete responses or partial responses as assessed by RECIST v1.1

SECONDARY OUTCOMES:
Best overall response (BOR) | 2.5 years
  BOR defined as the best response recorded from the date of T cell infusion until disease progression.
Time to response (TTR) | 2.5 years
  TTR defined as the duration between T cell infusion and the initial date of the confirmed response.
Duration of response (DoR) | 2.5 years
  DoR defined as the duration from the initial date of the confirmed response to the date of PD (or death).
Duration of stable disease (DoSD) | 2.5 years
  DoSD defined as the duration from the date of T cell infusion to the date of PD (or death).
Progression- free survival (PFS) | 2.5 years
  PFS defined as the interval between the date T cell infusion and the earliest date of disease progression based on RECIST v1.1 or death due to any cause.
Overall survival (OS) | 2.5 years
  OS defined the duration between T cell infusion and death due to any cause.
To evaluate the safety and tolerability of ADP-A2M4 with pembrolizumab by determining incidence of Adverse events (AEs) including serious adverse events (SAEs) | 2.5 years
  Determination of incidence, severity and duration of adverse events through assessment of adverse events including SAEs. Adverse events will be collected and graded as per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
To evaluate the safety and tolerability of ADP-A2M4 with pembrolizumab by determining the incidence, severity and duration of the AEs of special interest | 2.5 years
  Adverse events of special interest will be listed along with duration and toxicity grade.
To evaluate safety of ADP-A2M4 with pembrolizumab through measurement of Replication-competent Lentivirus in genetically engineered T-cells | 15 years
  Evaluation of RCL using PCR-based assay in peripheral blood.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - University of California San Diego, San Diego, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - Karmanos Cancer Insitute, Detroit, Michigan
  - Providence Cancer Institute Franz Head and Neck Clinic, Portland, Oregon
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - West Virginia University Cancer Institute, Morgantown, West Virginia